CLINICAL TRIAL: NCT02744846
Title: The Patient-Centered Outcomes Research Network (PCORnet) Obesity Observational Study: Short- and Long-Term Effects of Antibiotics on Childhood Growth
Brief Title: Short- and Long-Term Effects of Antibiotics on Childhood Growth
Acronym: ABX
Status: Completed | Type: Observational
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); National Patient-Centered Clinical Research Network (Other); ADVANCE CDRN (Unknown); Chicago Area Patient-Centered Outcomes Research Network (CAPriCORN) (Other); Greater Plains Collaborative Clinical Data Research Network (Other); Mid-South Clinical Data Research Network (Other); New York City Clinical Data Research Network (Other); OneFlorida Clinical Research Consortium (Other); PEDSnet: A Pediatric Learning Health System CDRN (Unknown); PORTAL CDRN (Unknown); Research Action for Health Network (REACHnet) (Other); Scalable Collaborative Infrastructure for a Learning Healthcare System (SCILHS) (Unknown); Genetic Alliance (Other); StatLog (Unknown)
Responsible Party: Principal Investigator, Jason Block, Assistant Professor, Harvard Pilgrim Health Care
Other Study IDs: OBS-1505-30699
Record Dates: First submitted 2016-04-13; First posted 2016-04-20 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Obesity
Keywords: antibiotics; children; pediatric; body mass index; Observational Study; Comparative Effectiveness Research; Obesity; Growth Trajectory; Cohort Study; Electronic Medical Record; Qualitative Research
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Children from birth to 5 years: Children from birth to 5 years where:
  1. 1 or more encounters with length and weight measured in the following age interval: 0-12 m, 12-30 m, and
  2. > 1 encounter with height and weight measured in either or both of the following age intervals: 4.0 to 5.9 y ("age 5 years"), or eligible to be followed to these ages for use in multiple imputation to account for missing data
  Interventions: Drug: Antibiotics exposure
- Children from birth to 10 years: Children from birth to 10 years where:
  1. 1 or more encounters with length and weight measured in each of the following age intervals: 0-12 m, 12-30 m, and
  2. > 1 encounter with height and weight measured in the following age interval: 9.0 to 10.9 y ("age 10 years"), or eligible to be followed to these ages for use in multiple imputation to account for missing data.
  Interventions: Drug: Antibiotics exposure

INTERVENTIONS:
Drug: Antibiotics exposure

SUMMARY:
The objectives of the proposed study are to assess the effects of different types, timing, and amount of antibiotic use in the first two years of life with (Specific Aim 1) body mass index (BMI) and obesity at ages 5 and 10 years and (Specific Aim 2) growth trajectories to age 5 years. In Specific Aim 3, the investigators will address how big the effects of antibiotics on obesity are within subgroups of the population, such as different racial/ethnic groups and whether the child's mother got antibiotics while she was pregnant.

The data for this study will come from electronic medical records of about 600,000 children from 42 healthcare systems within 10 Clinical Data Research Networks (CDRNs) across the United States. The investigators will get information on antibiotic prescribing in the first two years of life, then "virtually" follow these children to ages 5 and 10 years to see what their BMIs are, and how many of them are obese by clinical standards (i.e., body mass index exceeding the 95th percentile for age and sex).

In the main analyses, the CDRNs will not send any individual data to a central site. Rather, using sophisticated computer programs, the study's coordinating center will send "questions to the data," thus protecting the privacy of patients' and the healthcare systems' records. In some analyses, to check how well this "distributed research network" approach works, we will work with individual records whose identifying information has been stripped off ("de-identified data").

In our Secondary Aim, the investigators will employ focus groups of parents and in-depth interviews with clinicians to explore how best to put the findings into everyday practice.

Throughout the study, in addition to employing privacy-protecting approaches to analyzing and sharing data, the investigators will adhere to principles of inclusion, patient-centeredness, stakeholder engagement, effective governance, and protection of human subjects. At the end of the two-year project, the investigators will propose avenues for dissemination of the scientific findings and other products.

DETAILED DESCRIPTION:
Antibiotics are among the most valuable medical discoveries. Recent research on understanding of how bacteria in our gut use energy, however, raises concerns about whether broad-spectrum antibiotics, which are over-prescribed for mild infections, prescribed in early infancy may cause obesity during childhood. Obesity is a very common and serious condition among US children, particularly children from disadvantaged populations. Past studies examining the link between antibiotic use and childhood obesity are too small and they lack diversity as well as modern scientific tools to gauge the extent to which prescribing antibiotics can lead to excess weight gain. PCORnet, the National Patient-Centered Clinical Research Network, comprising very large networks of data from electronic medical records, provides an ideal test bed to address this question. Further, it is not clear how caregivers and clinicians will use the results of earlier studies to decide which antibiotics to prescribe when faced with common infections like ear infections.

Specific Aim 1: To evaluate the comparative effects of different types, timing, and amount of antibiotics used during the first two years of life on body mass index and risk of obesity at ages 5 (primary outcome age) and 10 (secondary) years. Hypothesis: There will be a "dose-response" relationship between the number of antibiotic courses given during the first 2 years of life and both higher BMI and the probability of obesity at ages 5 and 10 years. This relationship will be strongest for broad-spectrum antibiotics prescribed in the first 6 months of life.

Specific Aim 2: To assess the comparative effects of different types, timing, and amount of antibiotics used during the first two years of life on the rates and patterns of childhood growth during the first 5 years of life. Hypothesis: There will be a "dose-response" relationship between the number of antibiotic courses given during the first 2 years of life and subsequent growth trajectories of children in a pattern that increases children's risk of later overweight and obesity. This relationship will be strongest for broad-spectrum antibiotics prescribed in the first 6 months of life.

Specific Aim 3: To explore how the effects of different types, timing, and amount of antibiotics on childhood BMI, obesity risk and growth (Aims 1 and 2) vary according to patient socio-demographic, clinical, and maternal characteristics, including: 1) socio-demographic (Child sex, Child race/ethnicity, Geography, based on location of clinical facility); 2) Clinical (Prescription of medications that also cause obesity, esp. corticosteroids, Low birth weight or macrosomia in term infants); 3) Maternal for the subset of data partners listed in section B above that have linked maternal and child records (BMI, Maternal receipt of antibiotics during pregnancy, Type of delivery, i.e., Cesarean v. vaginal). Hypotheses: The antibiotic effects will not vary by socio-demographic or maternal characteristics. Long-term corticosteroid use will potentiate the effect of antibiotics on childhood obesity.

Secondary Aim: Through focus groups and in-depth interviews, to explore how parents and other caregivers and their providers assess information related to current and future benefits and risks, particularly for treatments such as antibiotics in early childhood, which can have substantial near-term benefits along with moderate long-term risks. The investigators will also explore how clinicians, health care organizations, and policy makers should best present study findings to help parents understand its strengths and limitations in the context of shared clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

1. 1 or more encounters with length and weight measured in each of the following age intervals: 0-12 months, 12-30 months, and
2. 1 or more encounters with height and weight measured after 24 months of age (need 1 or more measure at 4.0-5.9 years for the 5 year outcome and 1 or more measure at 9.0 to 10.9 years for the 10 year outcome), or eligible to be followed to these ages using multiple imputation to account for missing data.

Exclusion Criteria:

1. Biologically implausible length/height or weight measurements

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The study population will include children from age 0 to age 11 years. The population will be identified using data from participating sites formatted into the PCORnet Common Data Model (CDM).
Sampling Method: Probability Sample
Enrollment: 681739 (Actual)
Dates: Start 2016-02; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason P Block, MD, MPH, Principal Investigator — Harvard Pilgrim Health Care Institute; Christopher B Forrest, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia; Douglas Lunsford, Principal Investigator — Nationwide Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared publicly per Patient-Centered Outcomes Research Institute (PCORI) regulations 12 months after study completion. De-identified individual level data and aggregate data will be shared.

RESULTS

PARTICIPANT FLOW:
Groups:
- Children From Birth to 10 Years: Analysis Period 1:
  Children from birth to 5 years where:
  1. 1 or more encounters with length and weight measured in the following age interval: 0-12 m, 12-30 m, and
  2. >= 1 encounter with height and weight measured in the following age intervals: 4.0 to 5.9 y ("age 5 years")
  Analysis Period 2:
  Children from birth to 10 years where:
  1. Same criteria as above for the 5 year assessment, and
  2. >= 1 encounter with height and weight measured in the following age intervals: 9.0 to 10.9 y ("age 10 years")
Period: 5 Year Outcome Assessment
Arm/Group | Children From Birth to 10 Years
Started | 681739
Excluded Ineligible Patients | 319189 (Includes lost to follow-up and patients that had not reached age 4 years by end of study period)
Completed | 362550 (Number of patients that meet eligibility criteria)
Not Completed | 319189
Period: 10 Year Outcome Assessment
Arm/Group | Children From Birth to 10 Years
Started | 362550
Exclude Ineligible Patients | 305820 (Loss to follow-up, patients not yet 9 years, or systems that only had data from 2009 to 2016 or less)
Completed | 56730
Not Completed | 305820

BASELINE CHARACTERISTICS:
Groups:
- Children From Birth to 5 Years: Children from birth to 5 years where:
  1. 1 or more encounters with length and weight measured in the following age interval: 0-12 m, 12-30 m, and
  2. > 1 encounter with height and weight measured in either or both of the following age intervals: 4.0 to 5.9 y ("age 5 years"), or eligible to be followed to these ages for use in multiple imputation to account for missing data
  Antibiotics exposure
Arm/Group | Children From Birth to 5 Years
Number analyzed (Participants) | 681,739
Age, Customized [Count of Participants; unit: Participants]
  Less than 12 months | 681,739
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 324,864
  Male | 356,875
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 119,059
  Not Hispanic or Latino | 445,878
  Unknown or Not Reported | 116,802
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2,862
  Asian | 28,356
  Native Hawaiian or Other Pacific Islander | 2,930
  Black or African American | 170,007
  White | 363,759
  More than one race | 14,184
  Unknown or Not Reported | 99,641
Birth-related diagnoses [Count of Participants; unit: Participants]
  Prematurity | 52,752
  Heavy for gestational age newborn | 9,907
  Low birth weight | 5,828
  Macrosomia | 425
  No birth diagnosis | 612,827
Chronic conditions/categories [Count of Participants; unit: Participants]
  Asthma | 94,399
  Cardiovascular | 46,862
  Other congenital defect | 42,094
  Respiratory | 21,455
  Metabolic | 17,005
  Neuromuscular | 16,906
  Renal | 16,397
  Hematological/immunological | 14,547
  Endocrine | 6,602
  Malignant neoplasms | 6,593
  Gastrointestinal | 6,015
  No chronic condition diagnosis | 392,864

OUTCOME MEASURES:

1. Primary Outcome: Body Mass Index Z-score Difference at 48-72 Months, Exposed vs. No Antibiotics Less Than 24 Months
Description: BMI z-score measured between 48-72 months Body mass index z-scores are measures of relative weight adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Positive values below indicate a higher BMI z-score in children who received antibiotics versus those who did not.
Time Frame: 48-72 Months
Measure: Mean (95% Confidence Interval); unit: BMI z-score units
Groups:
- Children With no Complex Chronic Conditions; Children With Complex Chronic Conditions: Children from birth to 5 years where:
  1. 1 or more encounters with length and weight measured in the following age interval: 0-12 m, 12-30 m, and
  2. > 1 encounter with height and weight measured in the following age intervals: 4.0 to 5.9 y ("age 5 years"), or eligible to be followed to these ages for use in multiple imputation to account for missing data
  Antibiotics exposure
Arm/Group | Children With no Complex Chronic Conditions | Children With Complex Chronic Conditions
Number analyzed (Participants) | 310947 | 51603
BMI z-score units
  Any antibiotics vs. none <24 months of age | 0.04 [0.03 to 0.05] | 0.06 [0.04 to 0.09]
  Broad spectrum vs. none < 24 months of age | 0.04 [0.03 to 0.05] | 0.07 [0.05 to 0.10]
  Narrow spectrum vs. non <24 months of age | 0.02 [0.01 to 0.03] | 0.03 [-0.01 to 0.06]

2. Primary Outcome: Body Mass Index Z-score Difference at 10 Years, Exposed vs. No Antibiotics Less Than 24 Months
Description: BMI measured at 10 years Body mass index z-scores are measures of relative weight adjusted for child age and sex. The Z-score indicates the number of standard deviations away from a reference population in the same age range and with the same sex. A Z-score of 0 is equal to the mean. Positive values below indicate a higher BMI z-score in children who received antibiotics versus those who did not.
Time Frame: 10 years
Measure: Mean (95% Confidence Interval); unit: BMI z-score units
Groups:
- Children With no Complex Chronic Conditions; Children With Complex Chronic Conditions: Children from birth to 10 years where
  1. 1 or more encounters with length and weight measured in the following age interval: 0-12 m, 12-30 m, and
  2. > 1 encounter with height and weight measured in the following age interval: 9.0 to 10.9 y ("age 10 years"), or eligible to be followed to these ages for use in multiple imputation to account for missing data
Arm/Group | Children With no Complex Chronic Conditions | Children With Complex Chronic Conditions
Number analyzed (Participants) | 48785 | 7945
BMI z-score units
  Any antibiotics vs. none <24 months of age | 0.03 [0.01 to 0.06] | 0.09 [0.03 to 0.15]
  Broad spectrum vs. none < 24 months of age | 0.04 [0.01 to 0.06] | 0.08 [0.02 to 0.14]
  Narrow spectrum vs. non <24 months of age | 0.02 [-0.01 to 0.05] | 0.08 [-0.01 to 0.17]

ADVERSE EVENTS:
Time Frame: Not applicable - observational study only.
Description: Not applicable - observational study only.
Groups:
- Children From Birth to 10 Years: Children from birth to 10 years where:
  1. 1 or more encounters with length and weight measured in each of the following age intervals: 0-12 m, 12-30 m, and
  2. > 1 encounter with height and weight measured in the following age interval: 9.0 to 10.9 y ("age 10 years"), or eligible to be followed to these ages for use in multiple imputation to account for missing data.
  Antibiotics exposure
Arm/Group | Children From Birth to 5 Years | Children From Birth to 10 Years
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/46/NCT02744846/Prot_SAP_000.pdf